CLINICAL TRIAL: NCT02988648
Title: A Phase I/II Clinical Trial Evaluating the Safety and Clinical Activity of Radioiodide (131I-) as a Novel Targeted Therapy for Metastatic Breast Cancer That Overexpresses Functional Na/I Symporter
Brief Title: A Clinical Trial Evaluating the Safety and Clinical Activity of Radioiodide (131I-) as a Novel Targeted Therapy for Metastatic Breast Cancer That Overexpresses Functional Na/I Symporter
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was withdrawn due to lack of enrollment.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1607018035
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- radioiodide (I-) (Experimental): The Phase I portion will follow a 3+3 design with 4 dose levels (30, 60, 120, and 200 mCi) of I- treatment. The maximum tolerated dose (from Phase I) will be used in the Phase II efficacy assessment which will follow a Simon's optimal two-stage design.
  Interventions: Radiation: Radioiodide (131I-)

INTERVENTIONS:
Radiation: Radioiodide (131I-) — The Phase I portion will follow a 3+3 design with 4 dose levels (30, 60, 120, and 200 mCi) of I- treatment. The maximum tolerated dose (from Phase I) will be used in the Phase II efficacy assessment which will follow a Simon's optimal two-stage design.

SUMMARY:
The purpose of this phase I/II study is to evaluate the safety and clinical activity of Radioiodide (131I-) as a novel targeted therapy for metastatic breast cancer that overexpresses functional Na/I symporter. The study will enroll patients with metastatic breast cancer who have had clinical and/or radiographic evidence of disease progression on prior hormonal and/or chemotherapy.

DETAILED DESCRIPTION:
The primary objectives of the study are as follows:

1. To evaluate the feasibility of using 124I- PET/CT scans to identify patients whose metastatic lesions accumulate radioactive iodide and therefore are candidates for 131I- therapy.
2. Determine the frequency of iodide (124I) enriching metastatic breast cancer.
3. Evaluate the safety and clinical activity of one-time 131I treatment to patients who screen positive on 124I- PET/CT screening, positivity is defined as calculated iodide enrichment that will allow delivering 2000 cGy or more radiation to one or more metastatic lesion by administering up to 200mCi 131I-.

The secondary objectives of the study are as follows:

1. To investigate a correlation between NIS expression in tumor tissue with 124I- uptake on screening PET/CT scan

The Phase I portion will follow a 3+3 design with 4 dose levels (30, 60, 120, and 200 mCi) of I- treatment. The maximum tolerated dose will be used in the Phase II efficacy assessment which will follow a Simon's optimal two-stage design. The primary efficacy measure is objective tumor response rate (CR or PR) with targeted activity level of > 20% response rate.

The study will be terminated for futility if no tumor response is seen in the first 12 patients. If futility criteria is not met, a total of 37 eligible patients will be enrolled in the Phase II portion. If 4 or more responses are seen after 37 patients were evaluated, then the investigators will conclude that the regimen warrants further study.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all inclusion criteria in order to be considered for enrollment:

* Histologically confirmed breast cancer with clinical and/or radiological evidence of measurable or evaluable metastatic disease by Response Evaluation in Solid Tumors (RECIST) 1.1.
* Life expectancy ≥12 weeks.
* Radiologic or clinical evidence of disease progression on prior hormonal and/or chemotherapy
* There is no restriction on the number of prior lines of therapy.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of < 2.
* Full recovery to Grade ≤ 2 from any prior side effects of prior therapy for cancer including radiation therapy, chemotherapy, and/or immunotherapy.
* Adequate bone marrow function defined as white blood cells (WBCs) ≥ 3.0 × 109/L, neutrophils ≥ 1.5 × 109/L, platelets ≥ 100 × 109/L.
* Adequate renal function defined as serum creatinine < 1.5 mg/dL or creatinine clearance (GFR) > 40 mL/min calculated using the following formula: GFR = 175 x Serum Cr-1.154 x age-0.203 x 0.742 (female) and x 1.212 (if patient is African American).
* Adequate liver function defined as AST, ALT ≤ 3 × upper limit of normal (UNL) in the absence of liver metastasis and ≤ 5 × UNL with liver metastases; bilirubin < 1.5 × UNL; alkaline phosphatase ≤ 2.5 × UNL in the absence of liver metastasis and < 5 × UNL in case of bone metastases.
* TSH, T3 and free T4 must be within normal range.
* The patient should not have had intravenous or intrathecal iodinated contrast agents (IVP, CT with contrast, myelogram, angiogram) for 4 weeks prior to screening to their 124I- PET/CT scans and/or 131I- treatment.
* Patients with treated brain metastases are eligible if the brain metastases have remained stable for more than 4 weeks after completing therapy to the brain.
* Normal urine or serum Beta-HCG in premenopausal women of childbearing potential
* Women of childbearing potential must agree to use effective contraception during the treatment period and for at least 6 months after the last dose of 124I- and/or 131I- as these agents interfere with radioactive iodide uptake
* Signed informed consent.

Exclusion Criteria:

* Concurrent anti-tumor treatment including radiation therapy, hormonal and chemotherapy.
* Patients with symptomatic cardiac disease such as coronary artery disease, congestive heart failure, or atrial fibrillation.
* Significant gastrointestinal abnormalities, including: ulcerative colitis, chronic diarrhea associated with intestinal malabsorption, Crohn's disease, and prior surgical procedures affecting absorption.
* Women who are nursing or pregnant.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
objective tumor response rate | Up to 24 weeks
  The primary efficacy measure is objective tumor response rate (CR or PR) with targeted activity level of > 20% response rate.
  Patients should be followed regularly until disease progression and until resolution of all acute toxicities associated with treatment administration. If stable disease or resolution of toxicities takes longer than 24 weeks, follow up frequency will be determined by the treating physician.

CONTACTS AND LOCATIONS:
Overall Officials: Lajos Pusztai, M.D., D.Phil, Principal Investigator — Yale University: Professor of Medicine, Section of Medical Oncology
Locations (1):
- Smilow Cancer Center, New Haven, Connecticut, United States